CLINICAL TRIAL: NCT00878007
Title: Impact of Malaria Prevention on Health and Education in Kenyan Schoolchildren
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: World Bank (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 5503
Record Dates: First submitted 2009-04-07; First posted 2009-04-08 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Anaemia; Malaria
Keywords: Anaemia; Malaria; Literacy; Kenya
MeSH Terms: conditions — Anemia; Malaria; Literacy | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Intermittent screening and treatment (IST) for malaria.
  This intervention is a change from a previous intervention based on intermittent preventive treatment for malaria owning to the withdrawal of amodiaquine (one of the previous IPT drugs) in Kenya in 2009.
  Interventions: Drug: Intermittent screening and treatment for malaria
- 2 (Experimental): Enhanced teacher training on literacy instruction.
  Interventions: Behavioral: Teacher training on literacy instruction
- 3 (Experimental): Intermittent screening and treatment (IST) for malaria and enhanced teacher training on literacy instruction
  Interventions: Other: IST plus literacy instruction programme
- 4 (No Intervention)

INTERVENTIONS:
Drug: Intermittent screening and treatment for malaria — All children will be screened for malaria using rapid diagnostic tests (RDTs) once a term (thrice yearly). Children (with or without clinical malaria symptoms) found to be RDT-positive will be treated with artemether-lumefantrine according to national guidelines. Screening and treatment will be administered by district public health staff once a school term, observed by the evaluation research team.
  Arms: 1
Behavioral: Teacher training on literacy instruction — Education intervention designed to improved early grade literacy instruction, focusing on phonological awareness & vocabulary and relationship between letters and sounds in a systematic and explicit fashion. Specific interventions will include training on (i) how to monitor students' progress in large classes (ii) developing and using instructional materials for reading (iii) lesson planning for explicit teaching of letter-sound relationships (iv) instructional techniques for large classes.
  Arms: 2
Other: IST plus literacy instruction programme — Schools will receive both IST and the literacy instruction programme
  Arms: 3

SUMMARY:
While malaria represents one of the main health problems afflicting schoolchildren, the evidence base for policy development and programme implementation for school-based malaria control remains inadequate. A recent study in western Kenya showed that delivering intermittent preventive treatment (IPT) to schoolchildren improved rates of anaemia and classroom concentration, but did not improve school performance. This study aims to (i) investigate the impact of malaria prevention using a strategy of periodic screening using malaria rapid diagnostic tests and treatment positives using artemether-lumefantrine (AL) on health and education among schoolchildren and (ii) determine the interaction between health and improved literacy instruction. The study hypothesis is that that school-based malaria prevention will reduce rates of anaemia or improve educational outcomes in Kenyan schoolchildren, when compared to comparison schools. In addition, a programme of training for primary school teachers to improve literacy instruction will improve literacy rates and there will be no interaction between the malaria intervention and the education intervention, such that learning will not be improved when teaching is effective and children are healthy. The study will be undertaken in 101 randomly selected primary schools in Kwale District. The malaria intervention consists of screening all children using rapid diagnostic tests (RDTs) for malaria. Children (with or without clinical malaria symptoms) found to be RDT-positive will be treated with AL according to national guidelines. Screening and treatment will be administered by district public health staff once a school term, observed by the evaluation research team. This intervention has been changed from IPT due to the withdrawal of amodiaquine in Kenya. The education intervention includes a programme of training for primary school teachers to improve literacy instruction. The study is designed to detect a 25% reduction in anaemia and an improvement of 0.2 standard deviations in mathematics and literacy tests. Additional outcomes will also be measured including malaria parasitaemia, classroom attention and school attendance. Cost-effectiveness and community acceptability of the interventions will be assessed. Anaemia and educational outcomes will be assessed before interventions and 12 and 24 months later. Malaria parasitaemia using blood slides will only be assessed at follow-up.

DETAILED DESCRIPTION:
This study will be a factorial-design, cluster-randomised trial with a comparison group to assess the impact of (i) malaria prevention, based on screening and treatment, and (ii) enhanced literacy instruction by teachers on the health and educational achievement of healthy schoolchildren.

The target population in this study includes children attending primary schools in Kenya. The accessible population includes the children attending the participating primary schools in classes 1 and 5 in Kwale district. Schools will be randomized to one of four groups, receiving either the screening and treatment intervention alone, the education intervention alone, the malaria and education interventions combined, or neither intervention. The unit of analysis is the school, but individual-level analysis using suitable generalised linear models, adjusted for clustering by school, will also be undertaken to explore differences in impact of the interventions according to child age, sex, home environment, school quality as well as differences in the uptake of each intervention.

ELIGIBILITY:
Inclusion Criteria:

* Pupil enrolled at participating schools in classes 1 and 5;
* Provision of informed consent from parent or guardian;
* Provision of assent by student

Exclusion Criteria:

* Pupils unwilling to participate in the study;
* Known allergy or history of adverse reaction to study medications;
* Known or suspected sickle-cell trait

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5177 (Actual)
Dates: Start 2010-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Anaemia | 2 years
Education achievement assessed by a battery of tests of reading, writing and arithmetic | 2 years

SECONDARY OUTCOMES:
Prevalence of malaria parasitemia | 2 years
Concentration as assessed by classroom-based tests of sustained attention | 2 years
School attendance as assessed by class attendance registers | 2 years
Examination results as assessed by government examination scores | 2 years
Cost-effectiveness | 2 years
  Cost-effectiveness analysis will consider improvements in educational achievement and reductions in anaemia
Community acceptability | 2 years
  A modified stakeholder analysis will assess key people's views on the implementation and longer-term sustainability of the programme.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Brooker, DPhil, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- KEMRI-Wellcome Trust Programme, Nairobi, Kenya

REFERENCES:
- [Background] Brooker S, Okello G, Njagi K, Dubeck MM, Halliday KE, Inyega H, Jukes MC. Improving educational achievement and anaemia of school children: design of a cluster randomised trial of school-based malaria prevention and enhanced literacy instruction in Kenya. Trials. 2010 Oct 7;11:93. doi: 10.1186/1745-6215-11-93. PMID 20929566
- [Background] Okello G, Jones C, Bonareri M, Ndegwa SN, McHaro C, Kengo J, Kinyua K, Dubeck MM, Halliday KE, Jukes MC, Molyneux S, Brooker SJ. Challenges for consent and community engagement in the conduct of cluster randomized trial among school children in low income settings: experiences from Kenya. Trials. 2013 May 16;14:142. doi: 10.1186/1745-6215-14-142. PMID 23680181
- [Result] Halliday KE, Okello G, Turner EL, Njagi K, Mcharo C, Kengo J, Allen E, Dubeck MM, Jukes MC, Brooker SJ. Impact of intermittent screening and treatment for malaria among school children in Kenya: a cluster randomised trial. PLoS Med. 2014 Jan 28;11(1):e1001594. doi: 10.1371/journal.pmed.1001594. eCollection 2014 Jan. PMID 24492859
- [Result] Halliday KE, Karanja P, Turner EL, Okello G, Njagi K, Dubeck MM, Allen E, Jukes MC, Brooker SJ. Plasmodium falciparum, anaemia and cognitive and educational performance among school children in an area of moderate malaria transmission: baseline results of a cluster randomized trial on the coast of Kenya. Trop Med Int Health. 2012 May;17(5):532-49. doi: 10.1111/j.1365-3156.2012.02971.x. PMID 22950512
- [Result] Drake TL, Okello G, Njagi K, Halliday KE, Jukes MCh, Mangham L, Brooker S. Cost analysis of school-based intermittent screening and treatment of malaria in Kenya. Malar J. 2011 Sep 20;10:273. doi: 10.1186/1475-2875-10-273. PMID 21933376
- [Result] Okello G, Ndegwa SN, Halliday KE, Hanson K, Brooker SJ, Jones C. Local perceptions of intermittent screening and treatment for malaria in school children on the south coast of Kenya. Malar J. 2012 Jun 8;11:185. doi: 10.1186/1475-2875-11-185. PMID 22681850